CLINICAL TRIAL: NCT04201535
Title: Identification of Novel Molecular Targets for the Development of Therapies in Patients With Rheumatoid Arthritis Responsive to Disease-modifying Antirheumatic (DMARDs) But Wirh Progressive Bone Erosion (AREOS)
Brief Title: Identification of Novel Molecular Targets for Rheumatoid Arthritis Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: AREOS
Record Dates: First submitted 2019-12-05; First posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Arthritis, Rheumatoid; Bone Erosion
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1A:: at least 10 patients, maximum 70,with RA in remission, but presenting p• Group 1B: at least10 patients maximum 70, with RA in remission, without bone erosion A group of 80 controls,
  Interventions: Diagnostic Test: Protein arrays on plasma samples
- Group 2:: 10 patients with osteoarthritis (OA) who must undergo a surgical procedure.
  Interventions: Diagnostic Test: Protein arrays on plasma samples
- Group 3: 70 without RA and OA but hospitalized for any other orthopedics pathology who must undergo a surgical procedure.
  rogressive bone erosion who must undergo a surgical procedure.
  Interventions: Diagnostic Test: Protein arrays on plasma samples

INTERVENTIONS:
Diagnostic Test: Protein arrays on plasma samples — Protein arrays on plasma samples obtained from RA, OA patients and controls will be performed to identify a panel of acute phase proteins, cytokines and chemokines present at systemic levels and to highlight analogies and differences in the systemic protein profile.The synovial fluid will be used to identify through high-throughput MudPIT the proteins present in the synovial fluid of RA and OA patients.
  Other Names: Protein assay of the synovial fluid by high-throughput MudPIT

SUMMARY:
Aims of this study is to identify the mechanisms of the dissociation between the inflammatory activity and the joints destruction in patients with rheumatoid arthritis (RA) in remission but presenting a progression of the bone erosions.

160 total patients will be enrolled. Males and females RA patients in clinical remission or not, osteoarthritis patients and patients hospitalized for any other orthopedics pathology (used as controls) will be enrolled. From RA patients with bone erosion, OA patients and controls whole blood will be collected; from RA patients without bone erosion whole blood will be collected. From whole blood mononuclear cells will be isolated and plasma will be harvested. From both RA and OA patients synovial fluid will be collected along with mononuclear cells present in this fluid and from both RA and OA patients candidate for total articular replacement fragments of synovial membrane, cartilage, bone and bone marrow will be collected during surgery as waste material.

The nuclear cells isolated from whole blood, synovial fluid and bone marrow will be characterized using a panel of markers. Protein arrays on plasma samples obtained from RA, OA patients and controls will be performed to identify a panel of acute phase proteins, cytokines and chemokines present at systemic levels and to highlight analogies and differences in the systemic protein profile.

The synovial fluid will be used to identify the proteins present in the synovial fluid of RA and OA patients. The main identified target will be quantified and used as markers of erosion progression, to develop intra-articular pharmacological therapies and to suggest the therapeutic doses of drugs. The same kind of analysis will be performed even on tissues obtained from surgical patients (RA and OA patients) to establish the pathways involved and the tissue specific targets to be stimulated, i.e. with trophic factors, to promote the tissue homeostasis after switching-off the autoimmune and inflammatory processes.

DETAILED DESCRIPTION:
The general aim is to study the mechanisms of the dissociation between the inflammatory activity and the joints destruction in patients with rheumatoid arthritis (RA) in remission but presenting a progression of the bone erosions.

The primary aim is to detect differences between patients with AR in clinical remission, but presenting progressive articular erosion and patients in complete clinical and radiological remission, by characterizing the proteins, particularly the chromogranin A (CHGA), present both at articular and systemic levels.

The secondary aims are: to characterize the cellular inflammatory intra-articular infiltrate and the cells of the immune system present in the circulation; to characterize protein profile of the cells resident in the synovium, cartilage and bone of the damaged articulation. It is hypothesized that with this approach it is possible to detect protein or cellular markers able to identify early the patients at risk to progress towards articular erosion and to identify specific cellular and protein targets for the development of local or systemic therapies suitable for the control of the erosive RA.

This is a, observational with additional procedure, court, prospective study. 160 patients 80 RA patients (Group 1) of which:

* Group 1A: at least 10 patients, maximum 70,with RA in remission, but presenting progressive bone erosion who must undergo a surgical procedure.
* Group 1B: at least10 patients maximum 70, with RA in remission, without bone erosion A group of 80 controls,
* Group 2: 10 patients with osteoarthritis (OA) who must undergo a surgical procedure.
* Group 3:70 without RA and OA but hospitalized for any other orthopedics pathology who must undergo a surgical procedure.

Since several practical issues (e.g. unsuitableness or low amount of biological material) can occurs, we envision the possibility to recruit additional patients until the achievement of complete samples for the groups described.

Males and females RA patients in clinical remission or not, osteoarthritis patients and patients hospitalized for any other orthopedics pathology (used as controls) will be enrolled. For the RA patients, pharmacological treatment, laboratory data, RA activity, assessment of bone erosions with hands and feet x-ray will be recorded.

From RA patients with bone erosion, OA patients and controls whole blood will be collected; from RA patients without bone erosion whole blood will be collected. From whole blood mononuclear cells will be isolated and plasma will be harvested. A further tube will be collected for serum retrieval to perform CHGA dosage. From both RA and OA patients synovial fluid will be collected along with mononuclear cells present in this fluid and from both RA and OA patients candidate for total articular replacement fragments of synovial membrane, cartilage, bone and bone marrow will be collected during surgery as waste material.

The nuclear cells isolated from whole blood, synovial fluid and bone marrow will be characterized using a panel of markers indicated by the Human Immunology Project.

Protein arrays on plasma samples obtained from RA, OA patients and controls will be performed to identify a panel of acute phase proteins, cytokines and chemokines present at systemic levels and to highlight analogies and differences in the systemic protein profile.

The synovial fluid will be used to identify the proteins present in the synovial fluid of RA and OA patients. The main identified target will be quantified and used as markers of erosion progression, to develop intra-articular pharmacological therapies and to suggest the therapeutic doses of drugs. The same kind of analysis will be performed even on tissues obtained from surgical patients (RA and OA patients) to establish the pathways involved and the tissue specific targets to be stimulated, i.e. with trophic factors, to promote the tissue homeostasis after switching-off the autoimmune and inflammatory processes.

To reach this goal, the characterized protein profiles will be functionally evaluated by using Systems Biology techniques based on the study of protein-protein (PPI) interaction networks (8). Moreover, the protein profiles will be processed using statistics (Pearson, Spearman) able to evaluate the dependence between variables and to allow the building of protein co-expression networks (9). In both cases, PPI and/or co-expression networks, the study of the networks structure will allow the identification of hubs, bottlenecks and moduli (10) typical of the RA patients with or without erosion.

Serum will be sent to IRCCS Ospedale San Raffaele for the quantification of chromogranin A. Part of cells obtained from whole blood and synovial fluid will be sent to the IRCCS Ospedale pediatrico Bambino Gesù (Rome, Italy) for further immunological analysis.

ELIGIBILITY:
Inclusion Criteria:

* - patients with:

  1. rheumatoid arthritis treated with Disease-Modifying Antirheumatic Drugs (DMARDs), in remission but with progressive bone erosion who must undergo a surgical procedure (Group 1A).
  2. rheumatoid arthritis treated with DMARDs, in remission without bone erosion (Group 1B)
  3. osteoarthritis who must undergo a surgical procedure (Group 2).
  4. any other orthopedics pathology who must undergo a surgical procedure (Group 3).

     Exclusion Criteria:
* age < 18 or > 75 years old

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 160 patients 80 RA patients (Group 1) of which:
  * Group 1A: at least 10 patients, maximum 70,with RA in remission, but presenting progressive bone erosion who must undergo a surgical procedure.
  * Group 1B: at least10 patients maximum 70, with RA in remission, without bone erosion A group of 80 controls,
  * Group 2: 10 patients with osteoarthritis (OA) who must undergo a surgical procedure.
  * Group 3:70 without RA and OA but hospitalized for any other orthopedics pathology who must undergo a surgical procedure.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2017-12-21 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Protein analysis | 2nd year
  To detect differences between patients with AR in clinical remission, but presenting progressive articular erosion and patients in complete clinical and radiological remission, by characterizing:
  - the proteins, particularly the chromogranin A (CHGA), present both at articular and systemic levels.

SECONDARY OUTCOMES:
Inflammatory cell analysis | 2nd year
  To characterize the cells of the immune system present in the circulation and if possible the cellular inflammatory intra-articular infiltrate
Protein profile | 3rd year
  protein profile of the cells resident in the synovium, cartilage and bone of the damaged articulation

CONTACTS AND LOCATIONS:
Locations (1):
- Alessandra Colombini, Milan, Italy